CLINICAL TRIAL: NCT02343341
Title: Family-based Approach in a Minority Community Integrating Systems-Biology for Promotion of Health (FAMILIA)
Brief Title: Family-based Approach to Promotion of Health - FAMILIA (Project 1)
Acronym: FAMILIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GCO 14-0256 Project 1
Record Dates: First submitted 2015-01-15; First posted 2015-01-22 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Promoting Cardiovascular Health in Younger Age Group
Keywords: early childhood education; cardiovascular health; behavior change; community-based; family-based; prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preschool Health Promotion Education Program (Experimental): Children randomized to the intervention arm will receive a 4-month health promotion education program along with their parents/caregivers and teachers.
  Interventions: Behavioral: Preschool Health Promotion Education Program
- Control:Standard Curriculum (Other): The Standard curriculum control arm will receive the standard curriculum in their schools.
  Children randomized to the control arm will receive the health promotion education program for 4 months after the intervention arm has completed it
  Interventions: Behavioral: Preschool Health Promotion Education Program

INTERVENTIONS:
Behavioral: Preschool Health Promotion Education Program

SUMMARY:
Problem: Childhood obesity has more than doubled over the past 30 years, with nearly one-third of children aged 6 to 11 years being obese. These children are more likely to become obese adults and are at a higher risk for the development of diabetes, hypertension, heart disease and cancer.

Approach: This research tests the hypothesis that habits are formed very early in life and that children can help their parents live healthier lives. The investigators attempt to test this hypothesis by evaluating the impact of an educational program focusing on diet, physical activity, knowledge of the human body, and management of emotions for preschool children aged 3 to 5 years, their parents/caregivers and teachers. The investigators will first assess the environmental factors, facilitators, and barriers to implementation of a health promotion educational program tailored for preschoolers in Harlem, New York. This information will be used to tailor the educational program for the children in Harlem. The investigators will evaluate the effectiveness of the program in children aged 3 to 5 years by randomly assigning blocks of schools to a 4-month educational and playful health promotion intervention or to usual curriculum. The program will also have components for teachers and parents of these children in order to make their learning environment conducive to positive change. The impact of our program will be assessed on children's knowledge, attitudes, habits, weight, exercise and diet using simple questionnaires and measurements.

Impact: The investigators expect to demonstrate a positive impact on knowledge, attitudes and habits in preschool children in an under-served population. Also aim is to demonstrate that this early educational program can increase the proportion of preschool aged children with normal weight. This approach has the potential to meaningfully modify the projected rise in obesity and cardiovascular disease by affecting an entire generation of children. The investigators believe that the healthy habits that the children will acquire through this program will lead them to be healthier adults. Thus, the mission aligns closely with the American Heart Association's mission of, "Building healthier lives, free of cardiovascular diseases and stroke".

DETAILED DESCRIPTION:
Aim 1- Pilot: In the 1-year initial pilot period, the investigators will identify the contextual factors, facilitators and barriers that may impact the implementation of a preschool-based health promotion educational program in Harlem, using qualitative research methods: 1) focus group discussions among teachers; 2) focus group discussions among community leaders; and 3) focus group discussions among parents of preschool-aged children.

Subsidiary Aim 1.1: To use identified facilitators and barriers to develop a contextually and culturally appropriate model for a preschool-based health promotion educational program.

Subsidiary Aim 1.2: To implement a pilot intervention of the contextually and culturally adapted program at two preschools in Harlem. The investigators will assess for acceptability and feasibility, and make any necessary modifications prior to the implementation of the cluster-randomized trial.

Aim 2- Randomization: To evaluate the effectiveness of the preschool-based health promotion educational program on KAH-BEA: knowledge (K), attitudes (A), habits (H), BMI Z score (B), exercise (E) and Alimentation (A)(KAH-BEA) of approximately 600 preschool children, using a composite questionnaire-based score (KAH score) measuring the parameters related to the domains of diet, physical activity, health of the body and heart, and management of emotions, and weight and physical activity.

The investigators hypothesize that preschool children receiving the health promotion educational program will demonstrate a higher composite KAH score than controls.

The investigators hypothesize that a higher proportion of preschool children receiving the health promotion educational program will be eutrophic (B) than controls.

The investigators hypothesize that preschool children receiving the health promotion educational program will show higher levels of exercise and physical activity (E) and healthier diets (A) than controls.

For Aim 2, approximately 600 preschool children will be recruited from 15 schools in Harlem, NY, and perform a 3:2 (3 intervention: 2 control) cluster randomization of the schools. The preschool children will receive the intensive educational program for a period of four months. The primary assessments mentioned in Aim 2 will occur at approximately five months. At that time, the control schools will crossover to receive the educational program over the next four months.

Saliva will be collected from all children with assent. Saliva will be used to isolate DNA. The investigators will integrate this information with the one obtained from pre- and post-intervention blood adult samples to identify network models and predictors of primary prevention outcomes.

Aim 3-Sustainability: To evaluate the sustainability of the impact of a preschool-based health promotion educational program on the KAH-BEA of preschool children.

The investigators hypothesize the impact of an up to 4-month health promotion education program on the knowledge, attitudes, health, BMI, exercise level and diet of preschool children will be sustained out to 24 months.

For Aim 3, the preschool children will continue to be follow after all of them have received the educational intervention, up to approximately 24 months. The completion of this project will allow the assessment of effectiveness of multilevel approaches that intervene on children's environments and that aim to alter early life systems will prove to be effective in improving health habits in children and caregivers. The long-term expectation for these interventions is that they will reduce adolescent and adult obesity in these children and lead to improved CVD outcomes.

ELIGIBILITY:
Inclusion Criteria:

Fifteen preschools comparable in characteristics related to socio-economic level and ethnicity with the following criteria:

* The schools must be located in Harlem, NY;
* The schools must be public;
* The schools must have children 3, 4 and 5 years of age;
* The schools must provide meals for the children.
* The schools must make available use of their applicable program operation space.

Exclusion Criteria:

* Participation in any other major structured health intervention program similar to the FAMILIA Program during the evaluation of the program
* Inability to carry out all activities proposed by the FAMILIA Program

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 562 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Change in children's Knowledge, attitude, habit (KAH) scores | baseline and 5 months
  The mean change in KAH scores at immediate post-intervention (approximately 5 months) as compared to baseline.

SECONDARY OUTCOMES:
Change in children's BMI Z score, Exercise, and Alimentation (BEA) scores | baseline and 5 months
  The mean change in BEA scores at immediate post-intervention (approximately 5 months) as compared to baseline.
Change in children's Test of Emotion Comprehension scores | baseline and 5 months
  The mean change in BEA scores at immediate post-intervention (approximately 5 months) as compared to baseline.
Change in children's Knowledge, attitude, habit (KAH) scores | baseline and 24 months
  The mean change in children's Knowledge, attitude, habit (KAH) scores at approximately 24 months as compared to baseline.
Change in children's BMI Z score, Exercise, and Alimentation (BEA) scores | baseline and 24 months
  The mean change in BEA scores at approximately 24 months as compared to baseline.
Change in children's Test of Emotion Comprehension scores | baseline and 24 months
  The mean change in BEA scores at approximately 24 months as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (15):
- United States (15):
  - West Harlem Community Organization, Inc., New York, New York
  - East Harlem Community Organization, Inc., Site 2, New York, New York
  - East Harlem Council for Human Services, Inc., Site 1, New York, New York
  - Union Settlement Carver Childcare Center, New York, New York
  - Union Settlement Head Start at Franklin Plaza, New York, New York
  - Union Settlement Johnson, New York, New York
  - Union Settlement Leggett Memorial, New York, New York
  - Union Settlement Washington, New York, New York
  - Addie Mae Collins Head Start, Site 1, New York, New York
  - Addie Mae Collins Head Start, Site 2, New York, New York
  - Addie Mae Collins Head Start, Site 3, New York, New York
  - Association to Benefit Children Graham School, New York, New York
  - Lutheran Social Services, Site 11, New York, New York
  - Lutheran Social Services, Site 12, New York, New York
  - Lutheran Social Services, Site 14, New York, New York

REFERENCES:
- [Result] Vedanthan R, Bansilal S, Soto AV, Kovacic JC, Latina J, Jaslow R, Santana M, Gorga E, Kasarskis A, Hajjar R, Schadt EE, Bjorkegren JL, Fayad ZA, Fuster V. Family-Based Approaches to Cardiovascular Health Promotion. J Am Coll Cardiol. 2016 Apr 12;67(14):1725-37. doi: 10.1016/j.jacc.2016.01.036. PMID 27056780
- [Result] Bansilal S, Vedanthan R, Kovacic JC, Soto AV, Latina J, Bjorkegren JLM, Jaslow R, Santana M, Sartori S, Giannarelli C, Mani V, Hajjar R, Schadt E, Kasarskis A, Fayad ZA, Fuster V. Rationale and Design of Family-Based Approach in a Minority Community Integrating Systems-Biology for Promotion of Health (FAMILIA). Am Heart J. 2017 May;187:170-181. doi: 10.1016/j.ahj.2017.02.020. Epub 2017 Feb 22. PMID 28454800
- [Derived] Santos-Beneit G, Fernandez-Jimenez R, de Cos-Gandoy A, Bodega P, Diaz-Munoz R, Hill CA, Turco A, Santana M, Jaslow R, Peyra C, Carvajal I, Fuster V. Performance of Control Groups in Early Childhood Health Promotion Trials: Insights From the SI! Program. J Am Coll Cardiol. 2022 Aug 9;80(6):649-650. doi: 10.1016/j.jacc.2022.06.004. No abstract available. PMID 35926941
- [Derived] Fernandez-Jimenez R, Jaslow R, Bansilal S, Santana M, Diaz-Munoz R, Latina J, Soto AV, Vedanthan R, Al-Kazaz M, Giannarelli C, Kovacic JC, Bagiella E, Kasarskis A, Fayad ZA, Hajjar RJ, Fuster V. Child Health Promotion in Underserved Communities: The FAMILIA Trial. J Am Coll Cardiol. 2019 Apr 30;73(16):2011-2021. doi: 10.1016/j.jacc.2019.01.057. PMID 31023422